CLINICAL TRIAL: NCT02810457
Title: A Randomised, Parallel, Double Blinded Study to Compare the Efficacy and Safety of FKB238 to Avastin® In 1st Line Treatment for Patients With Advanced/Recurrent Non Squamous NSCLC in Combination of Paclitaxel and Carboplatin
Brief Title: Evaluation of FKB238 and Avastin in Patients With Advanced/Recurrent Non-squamous Non-small Cell Lung Cancer
Acronym: AVANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centus Biotherapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FKB238-002; 2015-004104-33 (EudraCT Number)
Record Dates: First submitted 2016-06-03; First posted 2016-06-23 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Cancer; Bevacizumab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FKB238 / paclitaxel / carboplatin (Experimental): Drug: FKB238:
  15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Drug: Paclitaxel:
  200 mg/m2 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Drug: Carboplatin:
  Area Under Curve (AUC) = 6.0 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Interventions: Drug: FKB238 (bevacizumab); Drug: Paclitaxel; Drug: Carboplatin
- Avastin / paclitaxel / carboplatin (Active Comparator): Drug: Avastin:
  15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Drug: Paclitaxel:
  200 mg/m2 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Drug: Carboplatin:
  AUC = 6.0 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Interventions: Drug: Avastin (bevacizumab); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: FKB238 (bevacizumab)
  Arms: FKB238 / paclitaxel / carboplatin
Drug: Avastin (bevacizumab)
  Arms: Avastin / paclitaxel / carboplatin
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
The purpose of this research study is to compare the effectiveness and safety of FKB238 against Avastin® in men and women with advanced/recurrent non squamous non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Newly diagnosed advanced (stage IV) /recurrent non-squamous NSCLC for which they had not received any systemic anti-cancer therapy for metastatic disease
* Histologically or cytologically confirmed diagnosis of predominantly non-squamous NSCLC
* Existence of at least 1 measurable lesion by RECIST v1.1
* Adequate hematological, renal and liver function
* Eastern Collaborative Oncology Group Performance Status (ECOG PS) 0 or 1
* Life expectancy longer than 6 months

Exclusion Criteria:

* Small cell lung cancer (SCLC) or combination SCLC and NSCLC. Squamous-cell tumors and mixed adenosquamous carcinomas of predominantly squamous nature
* Any unresolved toxicities from prior systemic therapy
* Known sensitizing epidermal growth factor receptor (EGFR) mutations or echinoderm microtubule-associated protein-like 4-anaplastic lymphoma kinase (EML4-ALK) translocation positive mutations
* Previous dosing with vascular endothelial growth factor (VEGF) inhibitor
* Known hypersensitivity to any excipients of the Investigational Products (IPs) and combination chemotherapy
* Use of prohibited concomitant medication
* Known Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) infection
* Fertile men or women of childbearing potential not using adequate contraception.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centus Biotherapeutics Limited, Study Director — Centus Biotherapeutics Limited
Locations (147):
- United States (11):
  - Research Site 7814 - Compassionate Care Research Group, Fountain Valley, California
  - Research Site 7811 - Innovative Clinical Research Institute, Whittier, California
  - Research Site 7803 - 21st Century Oncology, Jacksonville, Florida
  - Research Site 7812 - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Research Site 7810 - Edward H. Kaplan, MD and Associates, Skokie, Illinois
  - Research Site 7813 - Trinity Cancer Care Center, Minot, North Dakota
  - Research Site 7805 - Hematology & Oncology Associates, Inc., Canton, Ohio
  - Research Site 7801 - Gabrail Cancer Center, Canton, Ohio
  - Research Site 7804 - Tri-County Hematology & Oncology Associates, Inc., Massillon, Ohio
  - Research Site 7809 - Millennium Oncology, Houston, Texas
  - Research Site 7806 - Vista Oncology Inc. PS, Olympia, Washington
- Belarus (6):
  - Research Site 8507, Brest, Brest Oblast
  - Research Site 8505, Grodno, Hrodzenskaya Voblasts
  - Research Site 8501, Lyasny, Minsk Oblast
  - Research Site 8504, Minsk, Minsk Oblast
  - Research Site 8502, Mogilev, Mogilyov Oblast
  - Research Site 8506, Vitebsk, Vitebsk Oblast
- Bosnia and Herzegovina (6):
  - Research Site 8605, Tuzla, Tuzlanski Kanton
  - Research Site 8606, Banja Luka
  - Research Site 8602, Mostar
  - Research Site 8601, Sarajevo
  - Research Site 8603, Sarajevo
  - Research Site 8604, Zenica
- Bulgaria (2):
  - Research Site 0905, Sofia, Dobrich
  - Research Site 0904, Varna
- Croatia (3):
  - Research Site 1802, Zagreb, City of Zagreb
  - Research Site 1803, Zagreb, City of Zagreb
  - Research Site 1801, Osijek, Osjecko-baranjska Županija
- Georgia (5):
  - Research Site 2504, Batumi, Adjara
  - Research Site 2507, Kutaisi, Imereti
  - Research Site 2503, Tbilisi
  - Research Site 2505, Tbilisi
  - Research Site 2508, Tbilisi
- Germany (3):
  - Research Site 2605, Würselen, North Rhine-Westphalia
  - Research Site 2603, Kiel, Schleswig-Holstein
  - Research Site 2604, Hamburg
- Greece (3):
  - Research Site 3004, Athens
  - Research Site 3003, Thessaloniki
  - Research Site 3005, Thessaloniki
- Hungary (6):
  - Research Site 3303, Gyula, Bekes County
  - Research Site 3302, Deszk, Csongrád megye
  - Research Site 3301, Mátraháza, Heves County
  - Research Site 3305, Budapest
  - Research Site 3304, Budapest
  - Research Site 3306, Zalaegerszeg
- Italy (2):
  - Research Site 4107, Catania
  - Research Site 4106, Piacenza
- Japan (3):
  - Research Site 4301, Fukuyama-shi, Hiroshima
  - Research Site 4304, Kumamoto, Kumamoto
  - Research Site 4303, Sasebo-shi, Nagasaki
- Peru (4):
  - Research Site 5402, Arequipa
  - Research Site 5404, Arequipa
  - Research Site 5401, Lima
  - Research Site 5405, Lima
- Philippines (6):
  - Research Site 5505, Cebu City, Cebu
  - Research Site 5504, Makati City, National Capital Region
  - Research Site 5501, Manila, National Capital Region
  - Research Site 5502, Manila, National Capital Region
  - Research Site 5506, Manila, National Capital Region
  - Research Site 5503, Quezon
- Poland (7):
  - Research Site 5705, Toruniak, Kuyavian-Pomeranian Voivodeship
  - Research Site 5701, Krakow, Lesser Poland Voivodeship
  - Research Site 5708, Lodz, Lódzkie
  - Research Site 5702, Elblag, Warmian-Masurian Voivodeship
  - Research Site 5706, Olsztyn, Warmian-Masurian Voivodeship
  - Research Site 5711, Brzozów
  - Research Site 5703, Nowy Sącz
- Romania (7):
  - Research Site 6105, Cluj-Napoca, Cluj
  - Research Site 6106, Cluj-Napoca, Cluj
  - Research Site 6108, Floreşti, Cluj
  - Research Site 6101, Baia Mare
  - Research Site 6102, Constanța
  - Research Site 6103, Craiova
  - Research Site 6107, Iași
- Russia (27):
  - Research Site 6209, Arkhangelsk, Arkhangelskaya oblast
  - Research Site 6220, Ufa, Bashkortostan Republic
  - Research Site 6221, Belgorod, Belgorod Oblast
  - Research Site 6211, Chelyabinsk, Chelyabinsk Oblast
  - Research Site 6217, Kuzmolovskiy, Leningradskaya Oblast'
  - Research Site 6219, Saransk, Mordoviya, Respublika
  - Research Site 6225, Moscow, Moscow
  - Research Site 6203, Moscow, Moscow
  - Research Site 6230, Novgorod, Nizhny Novgorod Oblast
  - Research Site 6214, Novosibirsk, Novosibirsk Oblast
  - Research Site 6213, Novosibirsk, Novosibirsk Oblast
  - Research Site 6215, Omsk, Omsk Oblast
  - Research Site 6224, Omsk, Omsk Oblast
  - Research Site 6208, Orenburg, Orenburg Oblast
  - Research Site 6223, Rostov-on-Don, Rostov Oblast
  - Research Site 6205, Ryazan, Ryazan Oblast
  - Research Site 6234, Samara, Samara Oblast
  - Research Site 6235, Saint Petersburg, Sankt-Peterburg
  - Research Site 6212, Saint Petersburg, Sankt-Peterburg
  - Research Site 6216, Saint Petersburg, Sankt-Peterburg
  - Research Site 6202, Saint Petersburg, Sankt-Peterburg
  - Research Site 6210, Saint Petersburg, Sankt-Peterburg
  - Research Site 6201, Saint Petersburg, Sankt-Peterburg
  - Research Site 6229, Izhevsk, Udmurtiya Republic
  - Research Site 6228, Kursk
  - Research Site 6207, Magnitogorsk
  - Research Site 6222, Saint Petersburg
- Serbia (6):
  - Research Site 6401, Kamenitz, Vojvodina
  - Research Site 6402, Belgrade
  - Research Site 6403, Belgrade
  - Research Site 6404, Belgrade
  - Research Site 6405, Belgrade
  - Research Site 6406, Kragujevac, Šumadijski Okrug
- South Korea (4):
  - Research Site 6005, Busan, Busan Gwang'yeogsi
  - Research Site 6004, Suwon, Gyeonggido
  - Research Site 6002, Seoul, Seoul Teugbyeolsi
  - Research Site 6003, Ulsan, Ulsan Gwang'yeogsi
- Spain (8):
  - Research Site 7004, A Coruña, A Coruña
  - Research Site 7002, Castellon, Castellon
  - Research Site 7005, Córdoba, Córdoba
  - Research Site 7009, Jaén, Jaén
  - Research Site 7001, Burgos
  - Research Site 7007, Madrid
  - Research Site 7008, Murcia
  - Research Site 7003, Murcia
- Taiwan (4):
  - Research Site 7402, New Taipei City, Taipei
  - Research Site 7404, Douliu, Yunlin
  - Research Site 7403, Changhua
  - Research Site 7401, Taipei
- Thailand (7):
  - Research Site 7506, Bangkok, Bangkok
  - Research Site 7501, Hat Yai, Changwat Songkhla
  - Research Site 7504, Bangkok
  - Research Site 7507, Chiang Mai
  - Research Site 7505, Chiang Rai
  - Research Site 7503, Khon Kaen
  - Research Site 7502, Udon Thani
- Turkey (Türkiye) (4):
  - Research Site 7607, Ankara
  - Research Site 7605, Izmir
  - Research Site 7601, Izmir
  - Research Site 7606, Malatya
- Ukraine (10):
  - Research Site 7702, Chernivtsi, Chernivtsi Oblast
  - Research Site 7705, Kharkiv, Kharkivs’ka Oblast’
  - Research Site 7706, Odesa, Odesa Oblast
  - Research Site 7713, Lutsk, Volyn Oblast
  - Research Site 7707, Uzhhorod, Zakarpattia Oblast
  - Research Site 7709, Dnipro
  - Research Site 7701, Ivano-Frankivsk
  - Research Site 7708, Kryvyi Rih
  - Research Site 7704, Kyiv
  - Research Site 7710, Sumy
- Vietnam (3):
  - Research Site 8401, Hanoi, Ha Noi, Thu Do
  - Research Site 8402, Hanoi, Ha Noi, Thu Do
  - Research Site 8405, Hanoi, Ha Noi, Thu Do

REFERENCES:
- [Derived] Syrigos K, Abert I, Andric Z, Bondarenko IN, Dvorkin M, Galic K, Galiulin R, Kuchava V, Sriuranpong V, Trukhin D, Zhavrid E, Fu D, Kassalow LM, Jones S, Bashir Z; AVANA Investigators. Efficacy and Safety of Bevacizumab Biosimilar FKB238 Versus Originator Bevacizumab: Results from AVANA, a Phase III Trial in Patients with Non-Squamous Non-Small-Cell Lung Cancer (non-sq-NSCLC). BioDrugs. 2021 Jul;35(4):417-428. doi: 10.1007/s40259-021-00489-4. Epub 2021 Jul 15. PMID 34264503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening occurred at 146 centers in 24 countries (randomized at 136 centers, 24 countries) in Belarus, Bosnia & Herzegovina, Bulgaria, Croatia, Georgia, Germany, Greece, Hungary, Italy, Japan, South Korea, Peru, Philippines, Poland, Romania, Russia, Serbia, Spain, Taiwan, Thailand, Turkey, Ukraine, US and Vietnam. No screening occurred in Canada.
Pre-assignment Details: Of a total of 1023 patients who signed informed consent and were screened, 292 patients were not randomized. Of the 731 randomized patients, 2 patients were randomized in error and never received any study treatment, and 1 patient was randomized but withdrew consent prior to receiving any study treatment.
Groups:
- FKB238 / Paclitaxel / Carboplatin: Drug: FKB238:
  15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Drug: Paclitaxel:
  200 mg/m2 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Drug: Carboplatin:
  Area under the curve (AUC) = 6.0 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  FKB238 (bevacizumab)
  Paclitaxel
  Carboplatin
- Avastin / Paclitaxel / Carboplatin: Drug: Avastin:
  15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Drug: Paclitaxel:
  200 mg/m2 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Drug: Carboplatin:
  AUC = 6.0 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Avastin (bevacizumab)
  Paclitaxel
  Carboplatin
Period: Overall Study
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Started | 364 (362 patients received study treatment) | 367 (366 patients received study treatment)
Completed (Patients still in the study at DCO) | 37 | 38
Not Completed | 327 | 329
Not completed — Randomised but no treatment received | 2 | 1
Not completed — Objective PD assessed by RECIST v1.1 | 191 | 199
Not completed — Adverse Event | 37 | 43
Not completed — Patient decision | 31 | 35
Not completed — Patient lost to follow-up | 2 | 2
Not completed — Death | 39 | 28
Not completed — Ongoing at data cutoff and discontinued | 3 | 2
Not completed — Clinical progression | 15 | 16
Not completed — Investigator decision | 3 | 2
Not completed — Patient ineligibility | 3 | 0
Not completed — Miscalculated PD | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FKB238 / Paclitaxel / Carboplatin: Drug: FKB238:
  15 mg/kg IV infusion on Day 1 of each 21-day cycle.
  Drug: Paclitaxel:
  200 mg/m2 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  Drug: Carboplatin:
  AUC = 6.0 IV infusion on Day 1 of each 21-day cycle for at least 4 and no more than 6 cycles.
  FKB238 (bevacizumab)
  Paclitaxel
  Carboplatin
- Total: Total of all reporting groups
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin | Total
Number analyzed (Participants) | 364 | 367 | 731
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 238 | 224 | 462
  From 65-84 years | 126 | 143 | 269
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 129 | 248
  Male | 245 | 238 | 483
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 316 | 320 | 636
  Black and African American | 1 | 0 | 1
  Asian, other than Japanese | 37 | 37 | 74
  Japanese | 2 | 3 | 5
  American Indian or Alaska Native | 1 | 4 | 5
  Other | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Assessed as the Proportion of Patients With a Best Overall Response (BOR) of Either Complete Response (CR) or Partial Response (PR)
Description: The primary variable in this study was ORR, defined as the proportion of patients with a BOR of CR or PR (by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)). A BOR was defined as the best response (in the order of CR, PR, stable disease (SD), no evidence of disease (NED), progressive disease (PD), and not evaluable (NE)) among all post-baseline disease assessments that occurred until progression, or last evaluable assessment in the absence of progression prior to the initiation of subsequent anti-cancer therapy, irrespective of whether or not patients discontinued the study treatment. The 95% Pearson-Clopper confidence interval (CI) of ORR for each treatment arm was provided. Per RECIST v1.1 for target lesions and assessed by computed tomography (CT) or, if contraindicated, magnetic resonance imaging (MRI): CR=disappearance of all target lesions; PR=at least 30% decrease from baseline in the sum of diameters of target lesions. Overall Response=CR+PR.
Time Frame: Until data cut-off, which occurred 12 months after randomization of the last patient enrolled, for a total estimated period of time of up to approximately 30 months.
Population: In order to meet the Food and Drug Administration (FDA) requirement, the primary efficacy analysis of ORR was performed using the Intent-to-Treat (ITT) population (patients included in each treatment arm as randomized), and the blinded independent central review (BICR) radiological assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 364 | 367
percentage of participants | 51.6 [46.38 to 56.89] | 53.7 [48.43 to 58.87]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; Test type: Equivalence — A 90% CI for the ORR ratio between FKB238 and Avastin was estimated and compared to the margin (0.73 to 1.38), which was deemed to represent a clinically acceptable difference with respect to ORR. If the 90% CI was within the equivalence margin (0.73 to 1.38), an equivalence between FKB238 and Avastin, with respect to the ORR, was confirmed; Ratio in ORR = 0.96, 90% CI 2-sided [0.86 to 1.08]

2. Secondary Outcome: ORR at Week 19
Description: ORR (by RECIST v1.1) at Week 19 was defined as the proportion of patients with a BOR of CR or PR assessed at Week 19. Only tumor assessments performed up until 19 weeks (i.e. Week 18 assessment + 7 day assessment window) from randomization were considered in this analysis. Per RECIST v1.1 for target lesions and assessed by CT or, if contraindicated, MRI: CR=disappearance of all target lesions; PR=at least 30% decrease from baseline in the sum of diameters of target lesions. Overall Response=CR+PR.
Time Frame: From the date of randomization up to Week 19.
Population: In order to meet the FDA requirement, the secondary efficacy analysis of ORR was performed using the ITT population (patients included in each treatment arm as randomized), and the BICR radiological assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 364 | 367
percentage of participants | 47.8 [42.57 to 53.07] | 51.0 [45.71 to 56.18]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; Comparison between groups: Risk ratio in ORR at Week 19 by BICR; Test type: Other — Ratio in ORR analysis of FKB238 versus Avastin; Ratio in ORR = 0.94, 90% CI 2-sided [0.83 to 1.06]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: The event of interest for PFS was defined as the interval from the date of randomization until first documented disease progression or death from any cause, whichever occurs first. Disease progression was based on tumor assessments according to RECIST v1.1 criteria. The items of the overall response CR, PR, SD and NED were taken as progression-free whereas PD denoted disease progression. PFS was summarized using Kaplan-Meier estimates of the quartiles for each treatment arm, and 95% CIs for the medians were calculated. Per RECIST v1.1 for target lesions and assessed by CT or, if contraindicated, MRI: PD=at least a 20% increase in the sum of the longest diameter of target lesions, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: as for outcome 1
Population: This assessment was performed using the ITT population (patients included in each treatment arm as randomized) and the BICR radiological assessments.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 364 | 367
Months | 7.72 [7.46 to 7.98] | 7.62 [6.90 to 7.82]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; Hazard ratio and its 95% CI were calculated using the Cox regression model adjusting for baseline characteristics (randomization stratification factors, Eastern Cooperative Oncology Group (ECOG) performance status at baseline, gender, smoking history and age) with ties handled by the Efron method; Test type: Other — Hazard ratio analysis of FKB238 versus Avastin; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.82 to 1.16] — Treatment hazard ratio <1 favors FKB238

4. Secondary Outcome: Overall Survival (OS)
Description: The event of interest was defined as death from any cause. OS was defined as the interval from date of randomization until the date of death due to any cause. OS was summarized using Kaplan-Meier estimates of the quartiles for each treatment arm, and 95% CIs for the medians were calculated.
Time Frame: as for outcome 1
Population: This assessment was performed using the ITT population (patients included in each treatment arm as randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 364 | 367
Months | 14.13 [12.52 to 16.56] | 16.95 [14.65 to 19.02]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; Hazard ratio and its 95% CI were calculated using the Cox regression model adjusting for baseline characteristics (randomization stratification factors, ECOG performance status at baseline, gender, smoking history and age) with ties handled by the Efron method; Test type: Other — Hazard ratio analysis of FKB238 versus Avastin; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.96 to 1.45] — Treatment hazard ratio <1 favors FKB238

5. Secondary Outcome: Duration Of Response (DOR)
Description: DOR was evaluated in this study as a secondary efficacy endpoint. Only the patients defined as responders in the primary analysis of ORR were taken into account for the analysis of DOR. The event of interest was defined as first documented disease progression or death due to any reason, whichever occurred first. DOR was defined as the interval from the first documented response (as defined per RECIST v1.1) until the earlier date of the first documented disease progression or death due to any reason. The date of first documented response was taken as the date of the first tumor assessment with an overall visit response of CR or PR. Per RECIST v1.1 for target lesions and assessed by CT or, if contraindicated, MRI: CR=disappearance of all target lesions; PR=at least 30% decrease from baseline in the sum of diameters of target lesions. DOR was calculated in units of months.
Time Frame: as for outcome 1
Population: This assessment of DOR was based on patients with events in the ITT population (patients included in each treatment arm as randomized), and the BICR radiological assessments.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 188 | 197
months | 6.47 [5.39 to 7.69] | 6.31 [4.93 to 7.29]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; [analysis description as in outcome 4, analysis 1]; Test type: Other — Hazard ratio analysis of FKB238 versus Avastin; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.74 to 1.23] — Treatment hazard ratio <1 favors FKB238

6. Secondary Outcome: Disease Control Rate (DCR) Assessed as the Proportion of Patients With a BOR of Either CR, PR, SD or NED
Description: The DCR was defined as the proportion of patients defined as responders. The number and percentage of responders and non-responders and the 95% Pearson-Clopper CI of DCR for each treatment arm was provided. The odds ratio for treatment (FKB238 arm versus Avastin arm) and the corresponding 95% Wald CI were produced based on a logistic regression analysis of DCR. Per RECIST v1.1 for target lesions and assessed by CT or, if contraindicated, MRI: CR=disappearance of all target lesions; PR=at least 30% decrease from baseline in the sum of diameters of target lesions; SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study. DCR=CR+PR+SD (≥ 6 weeks).
Time Frame: as for outcome 1
Population: This assessment of DCR was based on patients in the ITT population (patients included in each treatment arm as randomized), and the BICR radiological assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 364 | 367
percentage of participants with response | 87.6 [83.81 to 90.84] | 87.5 [83.64 to 90.68]
Statistical Analysis 1: Comparison: FKB238 / Paclitaxel / Carboplatin vs Avastin / Paclitaxel / Carboplatin; The DCR was compared between treatment arms using logistic regression adjusting for baseline characteristics (randomization stratification factors, ECOG performance status at baseline, gender, smoking history and age); Test type: Other — Comparison between arms: Odds ratio; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.64 to 1.58] — Odds ratio >1 favors FKB238

7. Other Pre Specified Outcome: Serum Trough Concentration (Ctrough)
Description: Ctrough (pre-infusion) and serum maximum concentration (Cmax; at completion of infusion) were compared between treatment arms and time points, and descriptive statistics provided. Ctrough and Cmax concentrations were summarized using the pharmacokinetics (PK) population for each visit at which samples were taken. The pre-dose serum concentrations at Cycles 2, 4, and 6 were considered as Ctrough values and the post-dose serum concentrations at Cycles 1 and 4 were considered as Cmax values. PK data at Cycle 1 Day 1 pre-infusion were not calculable and are therefore not presented in the outcome measure data table. Data are only provided for the time points at which the serum trough concentration was measured.
Time Frame: Cycle 1 Day 1 (pre- and post-infusion), Cycle 2 Day 1 (pre), Cycle 4 Day 1 (pre and post), Cycle 6 Day 1 (pre), discontinuation visit, and every 12 weeks (up to 1 year [±14 days] after randomisation) until death, or the patient was lost to follow-up.
Population: All patients randomized to treatment who received at least 1 dose of investigational product with no important protocol deviations, and at least 1 serum drug concentration data after investigational product administration (PK population).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 345 | 351
ug/ml
  Cycle 1, Day 1 end of infusion: number analyzed (Participants) | 343 | 347
  Cycle 1, Day 1 end of infusion | 255.15 (184.3) | 245.11 (206.8)
  Cycle 2, Day 1 pre-infusion: number analyzed (Participants) | 325 | 327
  Cycle 2, Day 1 pre-infusion | 42.74 (91.9) | 48.48 (77.3)
  Cycle 4, Day 1 pre-infusion: number analyzed (Participants) | 280 | 284
  Cycle 4, Day 1 pre-infusion | 77.16 (69.4) | 83.26 (85.5)
  Cycle 4, Day 1 end of infusion: number analyzed (Participants) | 278 | 283
  Cycle 4, Day 1 end of infusion | 339.91 (91.3) | 373.92 (51.6)
  Cycle 6, Day 1 pre-infusion: number analyzed (Participants) | 247 | 253
  Cycle 6, Day 1 pre-infusion | 87.25 (124.5) | 108.22 (69.8)

8. Other Pre Specified Outcome: Proportion of Patients Developing Anti-drug Antibodies (ADAs)
Description: The ADA levels were summarized at baseline and post-baseline time points using descriptive statistics.
Time Frame: Pre-dose at Cycles 1, 2, 4 and 6, discontinuation visit, and every 12 weeks (up to 1 year [±14 days] after randomisation) until death, or the patient was lost to follow-up, whichever occurred first.
Population: Includes all patients randomized to treatment who received at least 1 dose of investigational product with no important protocol deviations, and who had non-missing baseline ADA and at least 1 non-missing post-baseline ADA result (ADA evaluable population).
Measure: Number; unit: percentage of participants
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
Number analyzed (Participants) | 305 | 305
percentage of participants
  ADA prevalence (ADA positive, baseline or post) | 3.0 | 3.0
  Treatment-emergent ADA positive (ADA incidence) | 2.3 | 2.3

9. Other Pre Specified Outcome: Adverse Events (AEs)
Time Frame: From the time of signature of informed consent, throughout the treatment period and up to and including the 30-days after the last dose of study treatment, for a total estimated period of time of up to approximately 30 months.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Vital Signs
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Hematology
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Clinical Chemistry
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Urinalysis
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Electrocardiogram
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Eastern Collaborative Oncology Group Performance Status
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Physical Examination
Time Frame: Up to approximately 30 days after last dose of study treatment.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent, throughout the treatment period and up to and including the 30-days after the last dose of study treatment, for a total estimated period of time of up to approximately 30 months. All ongoing and any new AEs/serious AEs (SAEs) identified during the 30 days after last dose were followed to resolution unless the event was considered by the investigator to be unlikely to resolve, or if the patient was lost to follow-up.
Description: All safety summaries and analyses were based on the Safety Population. Adverse events (AEs) were coded using the latest Medical Dictionary for Regulatory Activities(MedDRA) version (21.1). AEs were categorized as treatment-emergent AEs. Intensity of AEs was assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 grading system.
Arm/Group | FKB238 / Paclitaxel / Carboplatin | Avastin / Paclitaxel / Carboplatin
All-Cause Mortality (participants affected / at risk) | 195/362 | 177/366
Serious Adverse Events (participants affected / at risk) | 91/362 | 95/366
Other Adverse Events (participants affected / at risk) | 341/362 | 348/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB238 / Paclitaxel / Carboplatin (N=362) | Avastin / Paclitaxel / Carboplatin (N=366)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 9 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 18 (19)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 10 (12) | 9 (10)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (2)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FKB238 / Paclitaxel / Carboplatin (N=362) | Avastin / Paclitaxel / Carboplatin (N=366)
Hypertension (Vascular disorders) | 42 (47) | 44 (54)
Alanine aminotransferase increased (Investigations) | 38 (53) | 35 (45)
Aspartate aminotransferase (Investigations) | 32 (43) | 35 (45)
Blood alkaline phosphatase increased (Investigations) | 19 (24) | 27 (39)
Gamma-glutamyltransferase (Investigations) | 38 (48) | 31 (46)
Neutrophil count decreased (Investigations) | 24 (32) | 25 (30)
Platelet count decreased (Investigations) | 30 (48) | 25 (38)
Weight decreased (Investigations) | 41 (48) | 56 (62)
White blood cell count decreased (Investigations) | 24 (36) | 26 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 25 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 29 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 23 (36)
Anaemia (Blood and lymphatic system disorders) | 105 (135) | 119 (146)
Leukopenia (Blood and lymphatic system disorders) | 43 (58) | 50 (89)
Neutropenia (Blood and lymphatic system disorders) | 109 (163) | 145 (212)
Thrombocytopenia (Blood and lymphatic system disorders) | 44 (78) | 66 (102)
Headache (Nervous system disorders) | 18 (21) | 23 (24)
Neuropathy peripheral (Nervous system disorders) | 58 (63) | 52 (60)
Paraesthesia (Nervous system disorders) | 24 (26) | 22 (22)
Peripheral sensory neuropathy (Nervous system disorders) | 28 (28) | 25 (25)
Polyneuropathy (Nervous system disorders) | 16 (18) | 23 (31)
Asthenia (General disorders) | 37 (45) | 59 (71)
Fatigue (General disorders) | 41 (55) | 45 (48)
Non-cardiac chest pain (General disorders) | 18 (18) | 11 (15)
Pyrexia (General disorders) | 15 (17) | 21 (24)
Constipation (Gastrointestinal disorders) | 19 (23) | 21 (23)
Diarrhoea (Gastrointestinal disorders) | 35 (44) | 35 (41)
Nausea (Gastrointestinal disorders) | 52 (72) | 45 (57)
Vomiting (Gastrointestinal disorders) | 24 (29) | 18 (24)
Proteinuria (Renal and urinary disorders) | 24 (31) | 41 (52)
Alopecia (Skin and subcutaneous tissue disorders) | 154 (157) | 159 (162)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (49) | 36 (48)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (25) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (61) | 32 (73)
Decreased appetite (Metabolism and nutrition disorders) | 43 (56) | 42 (48)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (18) | 22 (29)
Pneumonia (Infections and infestations) | 18 (20) | 20 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publications/presentations made within 2 years of study completion require the Sponsor or CRO's prior written consent. The Sponsor shall be provided with copies of any materials relating to the study that they intend to publish/present at least 30 days in advance of publication, submission or presentation and the Institution shall withhold publication, submission or presentation for 90 days from the date on which the Sponsor receives the material (total time-frame of 120 days).

DOCUMENTS (2):
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02810457/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02810457/SAP_001.pdf